CLINICAL TRIAL: NCT03161184
Title: Evaluation of an mHealth Intervention to Improve Women's Access to Maternal Health Services in Rural Tanzania
Brief Title: Impact of a Smartphone Intervention on Tanzanian Women's Childbirth Location
Acronym: SUSTAIN1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: World Vision (Other); Muhimbili University of Health and Allied Sciences (Other)
Responsible Party: Principal Investigator, Daniel Sellen, Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 28832
Record Dates: First submitted 2017-05-01; First posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Maternal Death Affecting Fetus or Newborn; Delivery Complication; Obstetric Complication; Birth Injuries; Delivery; Injury, Maternal; Delivery Problem for Fetus
Keywords: maternal health; community health; health services; Tanzania; evaluation; cluster randomized trial
MeSH Terms: conditions — Birth Injuries; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Participants assigned to one of two groups in parallel for the duration of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (paper based) (Active Comparator): Women received prenatal household visits from CHWs who were trained on the Tanzania Ministry of Health and Social Welfare's National integrated Maternal, Newborn and Child Health (i-MNCH) paper-based protocols, i.e. received intervention "SUSTAIN Paperbased training of CHW (SOC)"
  Interventions: Behavioral: SUSTAIN Paperbased training of CHW (SOC)
- Intervention (Smart phone assisted) (Experimental): Women received prenatal household visits from CHWs trained on the following:
  A) National i-MNCH programme; and B) Smartphone-assisted counseling protocol: a smartphone application designed to assist with identification of danger signs during pregnancy, referral to health facilities, and MNCH counseling
  , i.e. received intervention "SUSTAIN Smartphone training of CHW (SP+)"
  Interventions: Behavioral: SUSTAIN Smartphone training of CHW (SP+); Behavioral: SUSTAIN Paperbased training of CHW (SOC)

INTERVENTIONS:
Behavioral: SUSTAIN Smartphone training of CHW (SP+) — Intervention (Smart phone assisted): During prenatal household visits, the smart phone based application guides CHW through electronic "decision tree" protocols, directing them to specific health/nutrition counseling topics and messages based on each woman's gestational age, and her answers to a specific series of diagnostic questions. Based on the client's gestational age, the tool directs CHW to lessons in an accompanying photo book, and reminds them to counsel on the importance of accessing timed and targeted maternal health services at health facilities. The application also assists CHW to identify danger signs during pregnancy, flags clients who require immediate referral to health facilities, and reminds CHW to follow-up with clients who were previously referred to clinics.
  Arms: Intervention (Smart phone assisted)
Behavioral: SUSTAIN Paperbased training of CHW (SOC) — SUSTAIN Paperbased training of CHW (SOC): During prenatal household visits, the CHW asks a specific series of diagnostic questions based on the client's gestational age, offers counsel on the importance of accessing appropriate maternal health services at health facilities and uses lessons in an accompanying photo book to deliver messages on a variety of maternal and newborn health and nutrition topics. CHW are trained to identify danger signs during pregnancy, flag clients who require immediate referral to health facilities, and follow-up with clients who were previously referred to clinics.

SUMMARY:
This study investigates whether training Community Health Workers (CHW) to use a smartphone-based prenatal counseling application as a "job aid" instead of the existing paper based standard is associated with increased women's use of maternal health services in Singida region, Tanzania.

DETAILED DESCRIPTION:
In low-income countries, frontline community health workers (CHWs) have potential to improve women's access to maternal health services through prenatal counseling and referral. However, CHW performance can often be enhanced with sufficient training, incentives, supportive supervision and job aids. Smartphone-based applications designed to assist CHWs with referrals, health education and client counseling may improve the quality of care delivered during household visits. There is a need for rigorous scientific studies on the impact of such interventions.

This study investigates whether CHWs' use of a smartphone-based application increases women's use of maternal health services in Singida region, Tanzania. It is hypothesized that smartphone-assisted counselling by CHWs can increase use of health facility-based delivery services compared to a control group of CHWs using standard paper-based protocols. This study is conducted within the context of larger project - SUSTAIN-MNCH Project (Supporting Systems to Improve Nutrition, Maternal, Newborn and Child Health), implemented by World Vision through multiple partners.

ELIGIBILITY:
Inclusion Criteria:

* client of one of the CHWs enrolled in the mHealth study
* visited at least once by a CHW following intervention (baseline training for CHWs) and during their most recent pregnancy
* most recent delivery was a live birth and the child is still living

Exclusion Criteria:

* None

Ages: 16 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity
Enrollment: 572 (Actual)
Dates: Start 2013-07-23 (Actual); Primary Completion 2014-06-25 (Actual); Study Completion 2014-06-25 (Actual)

PRIMARY OUTCOMES:
Delivery in a facility | Time between the participant's first prenatal visit by a trained CHW and the date of the postnatal household interview (up to 10 months)
  Participant delivered at or on the way to a health facility, measured by retrospective report at time of interview, after delivery
Antenatal care attendance | Time between the participant's first prenatal visit by a trained CHW and the date of the postnatal household interview (up to 10 months)
  Whether participant attended 4 ANC visits or more during their most recent pregnancy

SECONDARY OUTCOMES:
Gestational age at first contact/ANC | Time between the participant's first prenatal visit by a trained CHW and the date of the postnatal household interview (up to 10 months)
  Number of months into pregnancy the participant had first ANC visit
Iron supplementation during pregnancy | Time between the participant's first prenatal visit by a trained CHW and the date of the postnatal household interview (up to 10 months)
  Whether participant received 100 IFA tablets during pregnancy
HIV screening HIV Screening | Time between the participant's first prenatal visit by a trained CHW and the date of the postnatal household interview (up to 10 months)
  Whether the participant was screened for HIV during pregnancy
De-worming treatment during pregnancy | Time between the participant's first prenatal visit by a trained CHW and the date of the postnatal household interview (up to 10 months)
  Whether the participant reported during interview taking any listed de-worming medication during pregnancy
Bednet use | Time between the participant's first prenatal visit by a trained CHW and the date of the postnatal household interview (up to 10 months)
  Whether the participant slept under an insecticide treated bed net during pregnancy
Malaria prophylaxis during pregnancy | Time between the participant's first prenatal visit by a trained CHW and the date of the postnatal household interview (up to 10 months)
  Whether the participant reported during interview receiving two doses of IPTp during pregnancy
Tetanus Toxoid Vaccination | Time between the participant's first prenatal visit by a trained CHW and the date of the postnatal household interview (up to 10 months)
  Whether the participant received two TT vaccinations during pregnancy
Referrals | Time between the participant's first prenatal visit by a trained CHW and the date of the postnatal household interview (up to 10 months)
  Whether the participant was referred to a clinic during pregnancy by a CHW
Referral uptake | Time between the participant's first prenatal visit by a trained CHW and the date of the postnatal household interview (up to 10 months)
  Whether a referred participant went to the facility during pregnancy
Presence of partner at ANC | Time between the participant's first prenatal visit by a trained CHW and the date of the postnatal household interview (up to 10 months)
  Whether the participant's husband/spouse accompanied her to at least one ANC visit
Birth plan | Time between the participant's first prenatal visit by a trained CHW and the date of the postnatal household interview (up to 10 months)
  Whether the participant developed a birth plan during pregnancy
Early initiation of breastfeeding | Time between the participant's first prenatal visit by a trained CHW and the date of the postnatal household interview (up to 10 months)
  Whether the participant initiated breastfeeding within 1 hour after birth
Exclusive breastfeeding at 7 days | Time between the participant's first prenatal visit by a trained CHW and the date of the postnatal household interview (up to 10 months)
  Whether the participant breastfed exclusively for the first week after birth
BCG vaccination | Time between the participant's first prenatal visit by a trained CHW and the date of the postnatal household interview (up to 10 months)
  Whether the participant's child received BCG vaccination within the first week of life
Maternal knowledge of danger signs during pregnancy | Time between the participant's first prenatal visit by a trained CHW and the date of the postnatal household interview (up to 10 months)
  Number of pregnancy danger signs listed by participant

CONTACTS AND LOCATIONS:
Overall Officials: Daniel W Sellen, PhD, Principal Investigator — University of Toronto

IPD SHARING:
Plan to Share IPD: No
Sharing raw data is inconsistent with what was stated in the ethics application form and participant informed consent materials.

REFERENCES:
- [Derived] Hackett K, Lafleur C, Nyella P, Ginsburg O, Lou W, Sellen D. Impact of smartphone-assisted prenatal home visits on women's use of facility delivery: Results from a cluster-randomized trial in rural Tanzania. PLoS One. 2018 Jun 18;13(6):e0199400. doi: 10.1371/journal.pone.0199400. eCollection 2018. PMID 29912954